CLINICAL TRIAL: NCT02319031
Title: Open-Label, Randomized Study of Daclatasvir, Sofosbuvir, and Ribavirin for 12 vs. 16 Weeks in Treatment Naive and Treatment Experienced Patients With Genotype 3 Chronic Hepatitis C Infection Subjects With Compensated Advanced Fibrosis/Cirrhosis (F3/F4)
Brief Title: Safety and Efficacy Study of the Combination Daclatasvir (60 mg), Sofosbuvir (400 mg) and Ribavirin (Weight-based Dosing) for 12 or 16 Weeks in Subjects With Genotype 3 Chronic HCV Infection With or Without Prior Treatment Experience and Advanced Fibrosis or Compensated Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-326
Record Dates: First submitted 2014-12-12; First posted 2014-12-18 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1: Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) (Active Comparator): Oral dosing Daclatasvir 60mg once daily, Sofosbuvir 400mg once daily, and Ribavirin 1000-1200mg (weight based dosing) split into am and pm dosing
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir; Drug: Ribavirin
- Arm2 : Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks) (Active Comparator): Oral dosing Daclatasvir 60mg once daily, Sofosbuvir 400mg once daily, and Ribavirin 1000-1200mg (weight based dosing) split into am and pm dosing
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Daclatasvir
Drug: Sofosbuvir
Drug: Ribavirin

SUMMARY:
The purpose of the study is to determine if the combination of Daclatasvir, Sofosbuvir and Ribavirin for 12 or 16 weeks is safe and effective in the treatment of Genotype 3 Chronic Hepatitis C (HCV) in patients with advanced fibrosis or compensated cirrhosis. Patients in this study may have already been treated prior for HCV or may have never received treatment for their HCV.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must have Genotype 3 Chronic HCV
* Must have advanced fibrosis (F3) or compensated cirrhosis (F4)
* HCV RNA Viral load ≥ 10,000 IU/mL
* HCV Treatment naive or treatment-experienced

Exclusion Criteria:

* Non Genotype 3 or mixed genotypes
* Non advanced fibrosis or compensated cirrhosis
* Any prior treatment with NS5A inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol - Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- Australia (6):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Clayton, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Heidelberg, Victoria
- France (4):
  - Local Institution, Créteil
  - Local Institution, Grenoble
  - Local Institution, Paris
  - Local Institution, Vandœuvre-lès-Nancy

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- Available data/document: Primary Publication: PMID: 26822022 — http://www.ncbi.nlm.nih.gov/pubmed/26822022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 53 participants were enrolled. 50 participants were randomized and treated (24 to 12 week arm, 26 to 16 week arm). Reason for non-randomization was 3 no longer met study criteria.
Groups:
- Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks): Treatment-naïve and treatment-experienced participants with HCV Genotype 3 infection and advanced fibrosis or compensated cirrhosis (F3 or F4) were treated for 12 weeks with oral dosing of Daclatasvir (DCV) 60mg once daily, Sofosbuvir (SOF) 400mg once daily, and Ribavirin (RBV) 1000-1200mg (weight based dosing) split into am and pm dosing. Participants received either 400 mg (2 tablets for participants < 75 kg) or 600 mg (3 tablets for participants ≥ 75 kg) of RBV in the morning with food and 600 mg (3 tablets) of RBV in the evening with food. After the completion of the 12 week treatment period, participants were followed off treatment for 24 weeks. mg=milligram; kg=kilogram
- Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks): Treatment-naïve and treatment-experienced participants with HCV Genotype 3 infection and advanced fibrosis or compensated cirrhosis (F3 or F4) were treated for 16 weeks with oral dosing of Daclatasvir (DCV) 60mg once daily, Sofosbuvir (SOF) 400mg once daily, and Ribavirin (RBV) 1000-1200mg (weight based dosing) split into am and pm dosing. Participants received either 400 mg (2 tablets for participants < 75 kg) or 600 mg (3 tablets for participants ≥ 75 kg) of RBV in the morning with food and 600 mg (3 tablets) of RBV in the evening with food. After the completion of the 16 week treatment period, participants were followed off treatment for 24 weeks. mg=milligram; kg=kilogram
Period: Treatment Period
Arm/Group | Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) | Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks)
Started | 24 | 26
Completed | 23 | 26
Not Completed | 1 | 0
Not completed — Death | 1 | 0
Period: Follow-Up Period
Arm/Group | Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) | Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks)
Started | 23 | 26
Completed | 23 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Population: All enrolled participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) | Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks) | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (7.77) | 55.0 (5.75) | 54.1 (6.80)
Age, Customized [Number; unit: participants]
  <65 | 23 | 26 | 49
  >=65 | 1 | 0 | 1
Gender [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With a Sustained Virologic Response (SVR) at Follow-up Week 12 (SVR12)
Description: SVR12, defined as percentage of participants with hepatitis C virus (HCV) ribonucleic acid (RNA) < lower limit of quantitation (LLOQ), target detected (TD) or target not detected (TND) at follow-up Week 12. SVR12 imputation was based on Next Value Carried Backwards (NVCB) approach. HCV RNA measurements were excluded after the start of non-study anti-HCV medication on treatment or during follow-up.
Time Frame: Follow-up Week 12
Population: All treated participants: Enrolled participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) | Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks)
Number analyzed (Participants) | 24 | 26
percentage of participants | 87.5 [67.6 to 97.3] | 92.3 [74.9 to 99.1]

2. Secondary Outcome: Percent of Participants With a Sustained Virologic Response (SVR) at Follow-up Week 4 (SVR4) and Follow-up Week 24 (SVR24)
Description: SVR4, defined as percentage of participants with hepatitis C virus (HCV) ribonucleic acid (RNA) < lower limit of quantitation (LLOQ), target detected (TD) or target not detected (TND) at follow-up Week 4. SVR24, defined as percentage of participants with hepatitis C virus (HCV) ribonucleic acid (RNA) < lower limit of quantitation (LLOQ), target detected (TD) or target not detected (TND) at follow-up Week 24. SVR4 imputation was based on Next Value Carried Backwards (NVCB) approach. SVR24 imputation was based on missing being treated as non-responder. HCV RNA measurements were excluded after the start of non-study anti-HCV medication on treatment or during follow-up.
Time Frame: Follow-up Weeks 4 and 24
Population: All treated participants: Enrolled participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) | Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks)
Number analyzed (Participants) | 24 | 26
percentage of participants
  Follow-up Week 4 (SVR4) | 87.5 [67.6 to 97.3] | 96.2 [80.4 to 99.9]
  Follow-up Week 24 (SVR24) | 87.5 [67.6 to 97.3] | 92.3 [74.9 to 99.1]

3. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Discontinuation Due to Adverse Events (AEs), Grade 3 or Grade 4 (Grade 3/4) AEs, and Grade 3/4 Laboratory Abnormalities
Description: Serious adverse event (SAE) defined: a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Adverse event (AE) defined: any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. The degree of the adverse event or laboratory abnormality are evaluated by grades: Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death. Grading as per using National Cancer Institute Common Terminology Criteria (NCI CTC) Version 3.0 criteria.
Time Frame: Date of First Dose of Study Drug to 7 Days post last dose of study drug (up to 13 weeks or 17 weeks depending on the randomized treatment group)
Population: All treated participants: Enrolled participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) | Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks)
Number analyzed (Participants) | 24 | 26
participants
  Death | 1 | 0
  SAEs | 2 | 3
  Discontinuation due to AEs | 0 | 0
  Grade 3/4 AEs | 2 | 2
  Grade 3/4 Laboratory Abnormalities | 1 | 2

ADVERSE EVENTS:
Time Frame: SAEs were reported from date of first dose of study drug to 30 days post discontinuation of the last dose which was up to 16 weeks or 20 weeks depending on the randomized treatment group. Non-serious AEs were reported from date of first dose of study drug to 7 days post discontinuation of the last dose which was up to 13 weeks or 17 weeks depending on the randomized treatment group.
Description: Study initiated February 2015; study completed December 2015
Arm/Group | Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) | Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks)
Serious Adverse Events (participants affected / at risk) | 2/24 | 3/26
Other Adverse Events (participants affected / at risk) | 21/24 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) (N=24) | Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks) (N=26)
Arteriosclerosis (Vascular disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + Sofosbuvir + Ribavirin (12 Weeks) (N=24) | Daclatasvir + Sofosbuvir + Ribavirin (16 Weeks) (N=26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Headache (Nervous system disorders) | 7 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Irritability (Psychiatric disorders) | 5 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 6 | 7
Hypertension (Vascular disorders) | 0 | 3
Lethargy (Nervous system disorders) | 2 | 2
Asthenia (General disorders) | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.